CLINICAL TRIAL: NCT07016126
Title: D-BACE in Combination With Chemotherapy and Carelizumab for Resectable II-IIIA or Potentially Resectable T3-4N2 Stage IIIB NSCLC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY2024-1039-02
Record Dates: First submitted 2025-02-10; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2024-12

CONDITIONS: NSCLC (Non-small Cell Lung Cancer)
Keywords: Drug-eluting beads bronchial arterial chemoembolization
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- D-BACE in combination with chemotherapy and karelizumab (Experimental): 3 cycles of D-BACE (DCB-loaded microspheres loaded with epirubicin 50 mg) in combination with chemotherapy and karelizumab (the specific regimen of chemotherapy is determined by the investigator, and platinum-containing two-agent chemotherapy is generally used).
  Interventions: Combination Product: D-BACE in combination with chemotherapy and karelizumab

INTERVENTIONS:
Combination Product: D-BACE in combination with chemotherapy and karelizumab — 3 cycles of D-BACE (DCB-loaded microspheres loaded with epirubicin 50 mg) in combination with chemotherapy and karelizumab (the specific regimen of chemotherapy is determined by the investigator, and platinum-containing two-agent chemotherapy is generally used).

SUMMARY:
This study is a single-arm prospective single-center phase II study. Subjects are untreated resectable II-IIIIA or potentially resectable T3-4N2 stage IIIB NSCLC. 70 subjects will be enrolled in this prospective observation aimed at evaluating the clinical efficacy and safety of D-BACE in combination with neoadjuvant chemotherapy and carelizumab in patients with resectable II-IIIIA or potentially resectable T3-4N2 stage IIIB NSCLC. The treatment group regimen will be 3 cycles of D-BACE (DCB-loaded microspheres loaded with epirubicin 50 mg) in combination with chemotherapy and carelizumab (the specific regimen of chemotherapy will be determined by the investigator, and platinum-containing two-agent chemotherapy will generally be used). Adverse events will be monitored throughout the trial and graded for severity according to NCI CTCAE version 5.0. Tissue and blood specimens will be dynamically collected during the course of treatment for translational research.

DETAILED DESCRIPTION:
This study was a single-arm prospective single-center phase II study. Seventy patients with untreated resectable II-IIIA or potentially resectable T3-4N2 IIIB NSCLC will be included in this prospective study. The aim of this study is to evaluate the clinical efficacy and safety of D-BACE combined with neoadjuvant chemotherapy and camrelizumab in patients with resectable stage II-IIIA or potentially resectable T3-4N2 IIIB NSCLC. The treatment regimen was three cycles of D-BACE (epirubicin 50mg loaded on DCB microspheres) combined with chemotherapy and camrelizumab (the specific chemotherapy regimen was determined by the investigator, and generally platinum-based doubuse chemotherapy was used). Adverse events will be monitored throughout the trial and their severity will be graded according to the NCI CTCAE, version 5.0. At the same time, tissue and blood samples were dynamically collected during the treatment for related translational research exploration.

Patients could discontinue the regimen if:

Having comorbidities that significantly affect the assessment of clinical status or require discontinuation of protocol treatment (investigator's discretion); Unacceptable treatment toxicity; Disease recurrence or new primary invasive malignancy; At patient's request 4.1 Screening Subjects will complete whole-body PET-CT and contrast-enhanced brain MR Before enrollment to determine stage II-IIIB NSCLC. Patients were required to obtain adequate tissue or cell pathological diagnosis, relevant immunohistochemistry, PD-L1 protein immunohistochemistry and NGS testing before enrollment. At the same time, peripheral blood samples were collected before treatment for related indicators.

Tumor tissue was provided in newly obtained formalin-fixed specimens, preferably, or in old formalin-fixed paraffin-embedded specimens from sites not irradiated prior to biopsy. Tumor tissue must be archived (tissue blocks) before treatment. Slides ≤6 months old or recently fresh tumor biopsy slides submitted to the local study center),PD-L1 status determined:

PD-L1 positivity was defined as 1% tumor cell membrane staining positive in at least 100 evaluable tumor cells.

PD-L1 negative: defined as < 1% positive tumor cell membrane staining in at least 100 evaluable tumor cells PD-L1 nonevaluable/ambiguous: defined as subjects with insufficient sample quantity or quality to determine PD-L1 status by staining, or subjects with adequate tissue sample but still unable to determine PD-L1 status were classified together with PD-L1-negative subjects.

Screening (baseline) assessments were to be performed within 28 days before the first D-BACE.

4.2 Neoadjuvant therapy:

D-BACE should be administered within 28 days of baseline screening by:

One vial of 300-500μm DC Bead was loaded with 50mg epirubicin, and after full drug loading, 10-20ml of non-ionic contrast agent was added. Under the monitoring of digital subtraction angiography (DSA) equipment, femoral artery puncture was performed according to the technical specification of Seldinger puncture. Cobra, MIK, and single curved angiography catheters were used to explore the opening of tumor feeding arteries and perform angiography to understand the distribution of feeding arteries and tumor vessels. If systemic artery-pulmonary artery/pulmonary vein shunt is found during angiography, embolic materials such as blank microspheres, PVA or microcoils can be used to block the shunt. When the spinal artery was determined to be avoided, drug-loaded microspheres were injected into the tumor feeding artery through a microcatheter for chemoembolization. The injection rate was 1 mL/ min. The forward blood flow of the target embolized vessel must be maintained. "If" near blood stasis "is observed during the injection (i.e., the columnar contrast material in the vessel disappears after 2-5 heartbeats), the injection must be stopped to avoid backflow of the embolic agent, regardless of the actual amount of microspheres injected." In contrast, if "near blood stasis" did not occur after the target dose was fully infused, no additional bolusing of embolic agents was administered. After the operation, the arterial catheter and sheath were removed, the arterial puncture point was compressed and bandaged, and the hip joint was immobilized for more than 6 hours.

Neoadjuvant chemotherapy and camrelizumab should be administered within 7 days after D-BACE. The chemotherapy regimen was determined by the investigator. The chemotherapy regimen was generally platinum-based doubuse chemotherapy, such as pemetrexed (500mg/m2) plus carboplatin (AUC=5) (non-squamous carcinoma). Albumin paclitaxel (260mg/m2) combined with carboplatin (AUC=5).

4.3 Local treatment (surgery, SBRT, ablation, particle or D-BACE treatment) : PET-CT and contrast-enhanced MRI were performed after 3 cycles of D-BACE combined with chemotherapy and camrelizumab. The subsequent treatment strategy was evaluated by a multidisciplinary team. If surgical resection was considered, the specific surgical plan was determined by the surgeon. Accepted type of resection (negative margin), including lobectomy, sleeve lobectomy, bilateral lobectomy, or pneumonectomy; If the lesion could not be completely removed or the patient could not tolerate surgery after treatment, the radiotherapy department and interventional department would evaluate the treatment options such as local radiotherapy or ablation, seed, and D-BACE.

4.4 Adjuvant therapy after local treatment: For this study, adjuvant therapy after local treatment was determined by the investigator. The main regimens included standard 3-4 cycles of adjuvant chemotherapy or immunomaintenance therapy. EGFR mutations were deleted 4.5 Follow-up Each subject will be monitored for adverse events for at least 30 days after the end of treatment (serious adverse events will be collected for a maximum of 90 days after the end of treatment). Tumor assessments must continue according to the protocol and the subject will undergo post-treatment follow-up for disease status until one of the following events occurs :(1) disease progression; (2) initiation of non-investigational cancer treatment; (3) withdrawal of consent; (4) loss of follow-up or (5) death. Evaluation was performed by means of computed tomography (CT) of the chest and total abdomen (with enhanced venography, including the liver and adrenal glands and sites of suspected/known disease). Imaging evaluation was performed before each interventional embolization procedure. Postoperative baseline imaging was performed 3 months after local treatment and then every 12 weeks (±7 days) for up to 2 years, with primary chest (contrast-enhanced) CT. It is recommended to perform head MR At least once a year. If there are obvious neurological symptoms, head MR Should be performed in time.

4.6 Postoperative Radiotherapy Postoperative radiotherapy (PORT) will be administered at the discretion of the treating oncologist according to standard of care.

Based on the current international and domestic phase III randomized controlled trials of postoperative radiotherapy, postoperative adjuvant radiotherapy is not routinely performed for patients with complete resection, and for patients with non-R0 resection, postoperative adjuvant radiotherapy is not recommended.

4.7 Definition of end of study The start of the trial was defined as the first visit of the first subject. After 3 cycles of D-BACE combined with chemotherapy and camrelizumab, local intervention was performed within 6 weeks after assessment by imaging PET-CT and brain MRI enhancement scan, and subsequent adjuvant therapy was determined by the investigator. EGFR mutations were deleted. Survival follow-up continued for 5 years. The study was closed once survival follow-up was completed.

ELIGIBILITY:
Inclusion Criteria:

Only patients who met all the following criteria were eligible for inclusion in the study:

Provide written informed consent Male or female, aged 18-75 years Eastern Cooperative Oncology Group performance status ≤1 Measurable lesions in accordance with RECIST, version 1.1 Subjects must be able to provide a specimen containing tumor tissue or have a biopsy sample of newly resected tumor tissue available PD-L1 IHC testing was performed at a central laboratory during the screening phase

1. Before treatment, formalin-fixed, paraffin-embedded (FFPE) tissue blocks or non-stained tumor tissue sections and relevant pathology reports must be submitted for biomarker assessment. Tumor-tissue specimens could be fresh or archived within 6 months before enrollment.
2. The tissue must be core needle biopsy section, excisional biopsy section or open biopsy section;
3. It is recommended that fresh paraffin sections (PD-L1 assays be performed within 7 days of sectioning) slides be stored and transported in the dark
4. It is recommended that fresh tissue be fixed in 10% neutral buffered formalin for 24 to 48 hours The patient's lung function or other organ function was evaluated by the surgeon to tolerate local surgical treatment.

Adequate organ function assessment and laboratory screening should be performed within 7 days of initiation of therapy

Reproductive status:

1. A negative pregnancy test (serum or urine) in a woman of childbearing age within 72 hours before the start of treatment
2. women were non-lactating
3. For female patients, appropriate contraception should be used during treatment and for 6 months after the last dose of treatment (i.e., the time required for the 30-day ovulation cycle + the 5 half-lives of the drug).
4. Male subjects must agree to use appropriate contraception during treatment and for 7 months after the last dose of treatment (i.e., the duration of 90-day sperm turnover + 5 half-lives of the drug).

And male subjects had to be willing to avoid donating sperm during this period.

-

Exclusion Criteria:

Medical conditions Stage I, IIIB/IIIC (N3), and stage IV NSCLC patients with previous ICIs immunotherapy, targeted therapy, chemotherapy, and other systemic antitumor therapies were excluded.

Patients with allergy to contrast media were not eligible. Patients were excluded if their tumors had targeted alterations in EGFR and/or ALK or were known to have targeted alterations in ROS1, BRAF, HER-2, NTRK, MET, or RET. K-RAS mutations could be enrolled.

Active known or suspected autoimmune disease Participants were eligible if they had type I diabetes, hypothyroidism requiring only hormone-replacement therapy, skin conditions (e.g., vitiligo, psoriasis, or alopecia) that did not require systemic treatment, or other conditions that were not expected to recist in the absence of an external trigger.

Patients with active hepatitis B (positive hepatitis B surface antigen HBsAg test) or hepatitis C (positive HCV RNA test) Patients with previous HBV infection or a decommissioned HBV infection (defined as positive for the hepatitis B core antibody HBcAb and negative for HBsAg) were eligible to participate. Patients were required to provide HBV DNA test results before enrollment, and participants who were HBV carriers or required antiviral therapy were not eligible. Patients who tested positive for HCV antibodies could participate in the study only if they had negative PCR results for HCV RNA.

Any history of arterial thrombosis within 6 months of human immunodeficiency virus (HIV) -positive or acquired immunodeficiency syndrome (AIDS), History of deep vein thrombosis, pulmonary embolism, or any other major thromboembolism within 3 months uncontrolled angina, arrhythmia, or congestive heart failure within 5 years other active malignancy (except adequately treated carcinoma in situ of the cervix or basal cell or squamous cell skin cancer, superficial bladder cancer, or prostate cancer, breast cancer in situ) Patients with contraindications to local treatment (including surgery or intervention) as judged by the investigator.

Serious or uncontrolled medical illness The patient has psychosis or other medical conditions that result in treatment nonadherence History of severe hypersensitivity reactions to other monoclonal antibodies Patients who are unwilling to sign informed consent forms Patients who do not want follow-up Physical and laboratory tests Laboratory screening values must exclude the following criteria (CTCAE version 5 applies)

1. Bone marrow function:

   White blood cell count < 2000/uL, neutrophil < 1500/uL, platelet < 100×103/Ul, hemoglobin < 9.0g/dL
2. Liver function:

   1. Serum total bilirubin > 1.5 times the upper limit of normal value (ULN);
   2. In the case of liver metastases, AST and ALT were > 5×ULN and total bilirubin > 1.5ULN
3. Coagulation function:

   Abnormal coagulation function was defined as international normalized ratio (INR) or prothrombin time (PT) > 1.5 times ULN; If the subject was receiving anticoagulant therapy, PT was outside the intended use of anticoagulant drugs.
4. Renal function:

Urinary protein > 2+, or 24-hour urinary protein ≥1g; Serum creatinine > 1.5×ULN or calculated creatinine clearance (CrCl) < 50ml/min (using Cockcroft-Gault formula) Female CrCL=([140-age] × weight (kg) ×0.85)/(72× serum creatinine (mg/dL) Male CrCL=([140-age] × weight (kg) ×1.00)/(72× serum creatinine (mg/dL) Allergy and adverse drug reactions 1) A history of hypersensitivity to other monoclonal antibodies 2) A history of allergic or hypersensitive reactions to the components of the study drug Other exclusion criteria

1. Prisoners or subjects under compulsory confinement.
2. subjects who have been involuntarily detained for treatment of mental or physical illness (e.g., infectious disease).

Careful consideration has been given to the eligibility criteria for this study to ensure the safety of the study subjects and to ensure the availability of the study results.

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-12-22 (Actual); Primary Completion 2027-12-22 (Estimated); Study Completion 2027-12-22 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the pCR of resectable II-IIIA or potentially resectable T3-4N2 stage IIIB NSCLC treated with D-BACE in combination with chemotherapy and karelizumab | From enrollment to the end of treatment at 3 cycle (1 cycle is 21 day)
  Evaluation of the pathological complete response (pCR) of resectable II-IIIA or potentially resectable T3-4N2 stage IIIB NSCLC treated with D-BACE in combination with chemotherapy and karelizumab

SECONDARY OUTCOMES:
Evaluation of the MPR of resectable II-IIIA or potentially resectable T3-4N2 stage IIIB NSCLC treated with D-BACE in combination with chemotherapy and karelizumab | From enrollment to the end of treatment at 3 cycle (1 cycle is 21 day)
  Evaluation of the major pathological response (MPR) of resectable II-IIIA or potentially resectable T3-4N2 stage IIIB NSCLC treated with D-BACE in combination with chemotherapy and karelizumab
Evaluation of the ORR of resectable II-IIIA or potentially resectable T3-4N2 stage IIIB NSCLC treated with D-BACE in combination with chemotherapy and karelizumab | From enrollment to the end of treatment at 3 cycle (1 cycle is 21 day)
  Evaluation of the ORR of resectable II-IIIA or potentially resectable T3-4N2 stage IIIB NSCLC treated with D-BACE in combination with chemotherapy and karelizumab
Evaluation of the EFS of resectable II-IIIA or potentially resectable T3-4N2 stage IIIB NSCLC treated with D-BACE in combination with chemotherapy and karelizumab | From enrollment to the end of treatment at 3 cycle (1 cycle is 21 day)
  Evaluation of the EFS of resectable II-IIIA or potentially resectable T3-4N2 stage IIIB NSCLC treated with D-BACE in combination with chemotherapy and karelizumab
Evaluation of the PFS of resectable II-IIIA or potentially resectable T3-4N2 stage IIIB NSCLC treated with D-BACE in combination with chemotherapy and karelizumab | From enrollment to the end of treatment at 3 cycle (1 cycle is 21 day)
  Evaluation of the PFS of resectable II-IIIA or potentially resectable T3-4N2 stage IIIB NSCLC treated with D-BACE in combination with chemotherapy and karelizumab
Evaluation of the OS of resectable II-IIIA or potentially resectable T3-4N2 stage IIIB NSCLC treated with D-BACE in combination with chemotherapy and karelizumab | From enrollment to the end of treatment at 3 cycle (1 cycle is 21 day)
  Evaluation of the OS of resectable II-IIIA or potentially resectable T3-4N2 stage IIIB NSCLC treated with D-BACE in combination with chemotherapy and karelizumab
Evaluation as assessed by CTCAE v4.0 of the safety and tolerability of resectable II-IIIA or potentially resectable T3-4N2 stage IIIB NSCLC treated with D-BACE in combination with chemotherapy and karelizumab | From enrollment to the end of treatment at 3 cycle (1 cycle is 21 day)
  Evaluation as assessed by CTCAE v4.0 of the safety and tolerability of resectable II-IIIA or potentially resectable T3-4N2 stage IIIB NSCLC treated with D-BACE in combination with chemotherapy and karelizumab. Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

OTHER OUTCOMES:
Biomarkers (T-cell subsets) for predicting the efficacy (PFS and OS) of new D-BACE combined with chemotherapy and camrelizumab treatment and subsequent recurrence monitoring were explored | From enrollment to the end of treatment at 3 cycle (1 cycle is 21 day)
  Combined with the results of dynamic multi-omics exploratory analysis of individual patients, biomarkers (T-cell subsets) for predicting the efficacy of new D-BACE combined with chemotherapy and camrelizumab treatment and subsequent recurrence monitoring were explored.
The correlation of imaging response and pathological response with overall PFS and OS was observed and evaluated. | From enrollment to the end of treatment at 3 cycle (1 cycle is 21 day)
  The correlation of imaging response and pathological response with overall PFS and OS was observed and evaluated.
Changes in the infiltrating immune microenvironment | From enrollment to the end of treatment at 3 cycle (1 cycle is 21 day)
  The changes in the infiltrating immune microenvironment will be evaluated using flow cytometry and immunohistochemistry. Flow cytometry will be performed on peripheral blood samples to quantify the levels of various immune cell populations such as T cells, B cells, natural killer (NK) cells, and dendritic cells. Immunohistochemistry will be conducted on tissue samples to examine the spatial distribution and density of immune cells within the tumor microenvironment, including the expression of immune checkpoint proteins like programmed death-ligand 1 (PD-L1).

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong provincial people's hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest. Data or samples shared will be coded. Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact cuiwei@gdph.org.cn